CLINICAL TRIAL: NCT02344589
Title: The Effect of Local Anesthetic Volume Within the Adductor Canal on Quadriceps Function Evaluated by Electromyography: A Randomized, Observer-Masked, Placebo-Controlled Study in Volunteers.
Brief Title: The Effect of Local Anesthetic Volume Within the Adductor Canal on Quadriceps Function Evaluated by Electromyography
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ulrik Grevstad (Other)
Responsible Party: Sponsor-Investigator, Ulrik Grevstad, Associate professor, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SM-UG-14
Record Dates: First submitted 2015-01-16; First posted 2015-01-26 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Knee Arthroplasty, Total
Keywords: ACB; Adductor Canal Block; Peripheral Nerve Block
MeSH Terms: interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- ACB 10 (Experimental): ACB in right leg with 10ml of lidocaine 10mg/ml. Subject and assessor blinded, randomized. given on day 1, 2 or 3
  Interventions: Drug: Lidocaine
- ACB 20 (Experimental): ACB in right leg with 20ml of lidocaine 10mg/ml. Subject and assessor blinded, randomized. given on day 1, 2 or 3
  Interventions: Drug: Lidocaine
- ACB 30 (Experimental): ACB in right leg with 30ml of lidocaine 10mg/ml. Subject and assessor blinded, randomized. given on day 1, 2 or 3
  Interventions: Drug: Lidocaine
- FNB (Active Comparator): FNB in left leg with 20ml of lidocaine 10mg/ml on day 1. Unblinded arm, used for model control
  Interventions: Drug: Lidocaine
- Placebo (Placebo Comparator): ACB in left leg with 30ml of isotonic saline on day 2. Unblinded arm used for model control
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Lidocaine — used for the active blocks
  Other Names: lignocaine
  Arms: ACB 10; ACB 20; ACB 30; FNB
Drug: Saline — used for the placebo-block
  Other Names: NaCl
  Arms: Placebo

SUMMARY:
Our aim is to investigate which components of the quadriceps femoris muscle are affected following an ACB with different volumes (10, 20 and 30 ml) of 1% lignocaine evaluated by electromyography. Both a placebo treatment (20ml saline) and the femoral nerve block (20ml lignocaine 1%) as an active comparative will be used for model control. Further, we want to investigate the effect of volume on motor block. This will be evaluated by measuring the Maximum Voluntary Isometric Contraction (MVIC) of the quadriceps femoris muscle.

DETAILED DESCRIPTION:
The ACB has a well-proven analgesic effect after TKA, but we do not know which nerves that are affected by the block. Aside being a motor nerve, the nerve to the vastus medialis of the quadriceps femoris muscle, contains the second largest sensory contribution from the femoral nerve. It is probable that some of the analgesic effect of the ACB arises from blocking this nerve.

Even though the ACB is mainly a sensory nerve block, a study in healthy volunteers showed a small decline by 8% in quadriceps muscle strength(10). It is speculated that the decline in muscle strength was caused by the spread of local anesthetic to the nerve supplying the vastus medialis of the quadriceps femoris muscle. Three out of eleven of the volunteers experienced an even larger decline of 25 % in quadriceps muscle strength. It has been argued that this decline likely was caused by a proximal spread of the local anesthetic to the femoral triangle thereby resulting in an affection of the femoral nerve. In this study, a volume of 30 ml of local anesthetic was used.

We do not know the optimal volume for the ACB and we find it relevant to investigate to what extent and which parts of the quadriceps muscle gets affected when different volumes of a local anesthetic are injected into the adductor canal. Selective affection of the different components of the femoral quadriceps muscle can be assessed by non-invasive EMG recordings. Further, the quadriceps femoris muscle strength will be evaluated by measuring the MVIC following the different volumes. The EMG recordings will be voluntary (vEMG) measured during MVIC and stimulated (sEMG). sEMG is measured during transcutaneous electrical stimulation of the femoral nerve.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Subjects who gave their written informed consent to participating in the study after having fully understood the contents of the protocol and re-strictions.
* ASA 1
* Male
* BMI 18-30
* Physical exercise 1-3 hours/week

Exclusion Criteria:

* Subjects who cannot cooperate with the study.
* Subjects who cannot understand or speak Danish.
* Subjects with allergy to the medicines used in the study.
* Subjects suffering from alcohol and/or drug abuse - based on the investi-gator's opinion.
* Pathology or previous surgery or trauma to the lower limb.
* Intense exercise 24 h before the tests
* Intake of any analgesics 24 h prior to baseline measurements.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Difference between ACB-groups, one hour post-block, in amplitude of the rectified vEMG signal from the vastus medialis, expressed as percentage of the pre-block value. | one hour post-block
  vEMG=voluntary electromyography

SECONDARY OUTCOMES:
• Difference between ACB-groups, one hour post-block, in amplitude of the rectified vEMG signal from the vastus lateralis, expressed as percentage of the pre-block value. | one hour post block
  vEMG=voluntary electromyography
• Difference between groups, one hour post-block, in MVIC expressed as percentage of the pre-block value | one hour post-block
  MVIC=maximum voluntary isometric contraction. (Quadriceps femoris muscle)
• Difference between ACB-groups, one hour post-block, in amplitude of the rectified sEMG signal from the vastus medialis, expressed as percentage of the pre-block value. | one hour post-block
  sEMG= stimulated Electromyography
• Difference between ACB-groups, one hour post-block, in amplitude of the rectified sEMG signal from the vastus lateralis, expressed as percentage of the pre-block value. | one hour post-block
  sEMG= stimulated Electromyography
• Association between volume and MVIC. MVIC expressed as a percentage of the pre-block value. | one hour post-block
Difference in proportions between ACB-groups having an affection of both the saphenous nerve and the vastus medialis (but no other components of the quadriceps femoris muscle), one hour post block evaluated by EMG | one hour post-block
  For each subject a series of 5 voluntary EMG recordings during MVIC will be made to estab-lish the variability of the EMG recordings. This will be done prior to the blocks on each day resulting in 300 EMG recordings from the vastus medialis and 300 recordings from the vastus lateralis. From this variability we will establish a cut-off point (how large a decline in EMG amplitude is "synonymous" with affection of the nerve?). After the cut-off point has been established the EMG data will be presented in dichotomous form: affected/not affected

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Grevstad, MD, Principal Investigator — Gentofte Hospital
Locations (1):
- Rigshospitalet, Copenhagen, Denmark